CLINICAL TRIAL: NCT01292720
Title: Vitamin D Supplementation in Chronic Stable Heart Failure: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Vitamin D Supplementation in Chronic Stable Heart Failure
Acronym: VITD-HI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Karin Amrein, MD, Principal Investigator, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITD-HI
Record Dates: First submitted 2011-01-26; First posted 2011-02-09 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure; Vitamin D Deficiency
Keywords: vitamin D deficiency, vitamin D insufficiency, heart failure
MeSH Terms: conditions — Heart Failure; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (herbal oil)
  Interventions: Drug: Placebo
- Vitamin D (Experimental)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 90,000 IU followed by weekly 24,000 IU for 24 weeks of vitamin D3 (total dose: 666,000 IU)
  Other Names: Vitamin D
  Arms: Vitamin D
Drug: Placebo — Placebo in matching volumes
  Other Names: Herbal Oil
  Arms: Placebo

SUMMARY:
In cross-sectional and prospective cohort studies, vitamin D deficiency is associated with increased mortality, cardiovascular events including sudden cardiac death and stroke, diabetes, hypertension and impaired function of the immune and musculoskeletal system. The action of vitamin D on the cardiovascular system regulates cardiac function, endothelial and vascular smooth muscle, and, the renin-angiotensin system. Treatment with sufficiently high doses of vitamin D may represent a promising and inexpensive intervention option. To date, there are few data on the effect of cholecalciferol treatment in patients with chronic heart failure. The primary objective of this study is to investigate whether oral vitamin D supplementation improves chronic heart failure (measured with the surrogate parameter of NT-proBNP levels at month 0 and 6).

DETAILED DESCRIPTION:
A growing body of data suggests that low vitamin D levels may adversely affect cardiovascular health. For many cardiovascular events, seasonal variability with peak incidence in the winter months is proven. This may be attributable at least in part to declining body stores of vitamin D beginning with September. Recently, there have been several case reports about severe cardiomyopathy caused by vitamin D deficiency, especially in dark-skinned children who had low vitamin D levels. The heart is an important target organ for vitamin D, both on a genomic and nongenomic level. Myocytes express the vitamin D receptor and several models of hypertension in animal studies have shown that vitamin D treatment is able to prevent cardiac hypertrophy [9-10]. Vitamin D seems to inhibit activation of the cardiac renin-angiotensin system as well as the expression of genes involved in the development of myocardial hypertrophy. There is accumulating evidence that vitamin D deficiency may be an important factor in the development of congestive heart failure and sudden cardiac death.

In chronic hemodialysis patients, vitamin D supplementation has been associated with reduction of cardiac hypertrophy and a reduction of QT dispersion, the latter being considered a major risk factor for sudden cardiac death. A small study from 1984 showed an improvement in left ventricular function after treatment with cholecalciferol in hemodialysis patients. A recent study from our group has reported a negative correlation of 25(OH)D levels with NT-pro-BNP levels, New York Heart Association functional classes and impaired left ventricular function. Furthermore, hazard ratios for death attributable to heart failure and sudden cardiac death were 2.84 and 5.05, respectively, when patients with 25(OH)D <25ng/ml were compared with those having serum levels of 25(OH)D >75 ng/ml [11]. The anti-inflammatory properties of vitamin D also appear to play a role in congestive heart failure, as studied in a recent interventional trial. In animal models, vitamin D deficiency was proven to be associated with developing myocardial hypertrophy and fibrosis with aberrant cardiac contractility and relaxation. Moreover, vitamin D deficiency can raise parathyroid hormone secretion, which in turn may increase insulin resistance and be associated with the development of diabetes, hypertension and inflammation. In summary, vitamin D seems to exert a multitude of different effects all working in concert to protect the vascular and cardiac system by influencing various hierarchical levels of biologic response.

Recently, a randomized controlled trial in a subgroup of patients with heart failure(n=105, ≥ 70 years) was able to demonstrate a significant decrease in BNP levels at 10 and 20 weeks, while the primary endpoint "functional capacity" and quality of life did not differ between intervention and placebo group.

Because in this latter trial, even the intervention group did not reach normal vitamin D levels, we will use a higher dose of vitamin D given in shorter intervals.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable heart failure (NYHA II-IV, ejection fraction ≤ 40%)
* ≥ 45 years
* 25 (OH) Vitamin D ≤ 30ng/ml

Exclusion Criteria:

* hypercalcemia (total serum calcium > 2.65 mmol/l OR ionized calcium > 1.35 mmol/l)
* nephro-/urolithiasis (≤1 year)
* known granulomatous diseases (active tuberculosis, sarcoidosis)
* pregnancy

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
NT-pro BNP | month 0, 6
  Change from Baseline in NT-pro BNP serum level at 6 months

SECONDARY OUTCOMES:
Percentage of patients with 25(OH)D ≥ 30 ng/ml at month 6 | 6 months
  Percentage of patients with 25(OH)D ≥ 30 ng/ml at month 6
Serum calcium | month 0, 6
  Serum calcium levels
DXA | month 0,12
  Dual energy X-ray absorptiometry including body composition at month 0 and 12 (alternatively month 6)
Urinary calcium | month 0,6
  Urinary calcium (spot urine)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Amrein, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria